CLINICAL TRIAL: NCT00985920
Title: Efficacy of Intraoperative Topical Application of Tranexamic Acid in Reducing Perioperative Bleeding in Total Knee Arthroplasty
Brief Title: Topical Tranexamic Acid for Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Dr. Jean Wong, Staff Anesthesiologist , Assistant Professor, Anesthesia Department, Toronto Western Hospital, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 070199A
Record Dates: First submitted 2009-09-28; First posted 2009-09-29 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Surgical Blood Loss; Total Knee Arthroplasty
Keywords: blood loss; postoperative
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tranexamic acid, 1.5 g (Experimental): 1.5 g of tranexamic acid in 50 cc of normal saline solution is given to the patients.
  Interventions: Drug: tranexamic acid
- Tranexamic acid, 3.0 g (Experimental): 3.0 g of tranexamic acid in 50 cc of normal saline is given to the patients.
  Interventions: Drug: tranexamic acid
- Placebo, saline (Placebo Comparator): 50 cc of sterile normal saline solution is given to the patients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tranexamic acid — Patients will receive a solution containing either 1.5g or 3 g of tranexamic acid in 50 ml of normal saline (0.9% sodium chloride) or only 50 ml of saline without TA (placebo).
  The treatment solution will be prepared under sterile conditions and coded at TWH pharmacy. In the OR the sterile bag containing the solution will be given to the scrub nurse. The contents (50 ml) will be emptied in a sterile surgical bowl. TA or placebo solution (50 ml) will be then applied to the open joint and tissues by the bulb syringe and will be left in contact with the tissues for 5 minutes. Excess solution will be subsequently suctioned by placing the suction tip on the cemented component without touching the joint and surrounding tissues.
  Other Names: cyklokapron
  Arms: Tranexamic acid, 1.5 g; Tranexamic acid, 3.0 g
Drug: Placebo — Patients will receive a solution containing either 1.5g or 3 g of tranexamic acid in 50 ml of normal saline (0.9% sodium chloride) or only 50 ml of saline without TA (placebo).
  The treatment solution will be prepared under sterile conditions and coded at TWH pharmacy. In the OR the sterile bag containing the solution will be given to the scrub nurse. The contents (50 ml) will be emptied in a sterile surgical bowl. TA or placebo solution (50 ml) will be then applied to the open joint and tissues by the bulb syringe and will be left in contact with the tissues for 5 minutes. Excess solution will be subsequently suctioned by placing the suction tip on the cemented component without touching the joint and surrounding tissues.
  Other Names: normal saline
  Arms: Placebo, saline

SUMMARY:
Total knee arthroplasty (TKA), the definitive treatment of osteoarthritis, is often associated with excessive postoperative bleeding due to increased fibrinolysis. Hence, the objective of the proposed study is to determine the role of topical application of tranexamic acid (TA), an anti-fibrinolytic agent, into the knee joint just before closure during TKA to reduce perioperative bleeding. The investigators' hypothesis is that in patients undergoing unilateral primary TKA, intraoperative application of 1.5 g or 3.0g topical TA into the knee joint before closure reduces perioperative bleeding as depicted by a decrement in the maximal drop in hemoglobin concentration following surgery. This proposal describes a randomized, double-blinded, placebo-controlled clinical trial with three arms. The primary outcome is the extent of the postoperative reduction in hemoglobin levels. Secondary outcomes will include transfusion requirements, hospital stay, joint functionality, quality of life and safety of using topical TA. Topical application of TA is a novel intraoperative approach that has not been used or studied in TKA. However if it is effective, it will directly reduce postoperative intra-articular bleeding without subsequent systemic absorption and thromboembolism. In addition, the reduction in microvascular intra-articular bleeding will lead to less pain and infection rates as well as improved surgical functional outcomes.

DETAILED DESCRIPTION:
Three million (1 in 10) Canadians suffer from Osteoarthritis (OA). Total knee arthroplasty (TKA), i.e. knee replacement surgery is the definitive treatment for knee osteoarthritis which alleviates pain and restores physical functioning. However, it can be associated with excessive postoperative bleeding leading to increased mortality and morbidity. The current blood conservation techniques, i.e. preoperative erythropoietin and autologous blood donation, do not reduce bleeding from the surgical site. As a result, many patients require blood transfusion with the associated risks and costs. In TKA, postoperative bleeding is attributed to diffuse microvascular bleeding as a result of increased fibrinolytic activity caused by releasing of the tourniquet which is routinely applied to provide appropriate surgical exposure during surgery. Therefore, tranexamic acid (TA), an antifibrinolytic agent which blocks the dissolution of hemostatic fibrin, can decrease blood loss following TKA. The systemic administration of TA, however, carries the risk of thromboembolic events such as deep vein thrombosis (DVT) or pulmonary embolism (PE). In TKA, this is of greater importance, as the patients are at higher risk of thromboembolic events. Topical application of TA in the surgical field is a cost-effective and simple route of administration that has been shown to reduce bleeding in dental, cardiac, and spine surgeries while minimizing systemic absorption and thromboembolism. Another major advantage of this approach is to prevent diffuse microvascular bleeding at the site of raw tissue surfaces resulting in decreased infection rate, pain, and increased range of motion (ROM) of the knee joints. In spite of these potential benefits, the innovative idea of topical application of TA has not been studied in TKA. However, if it is shown to be efficacious in decreasing postoperative bleeding, it can be incorporated into routine clinical practice with immediate beneficial impacts on patient care and quality of life.

Hypothesis:

In patients undergoing unilateral primary/revision TKA, intraoperative application of 1.5 g or 3 g topical TA into the surgical wound for five minutes before closure reduces perioperative bleeding as depicted by the maximal drop in systemic hemoglobin concentration during the postoperative period.

General Objective:

To study the role of tranexamic acid as a therapeutic tool, applied intraoperatively into the surgical wound, to reduce perioperative blood loss in patients undergoing a unilateral primary/revision TKA.

Specific Objectives:

To determine:

* the efficacy of topical application of TA to reduce perioperative transfusion requirements.
* the safety of topical application of TA (complications such as DVT).
* the systemic absorption of TA after topical application into the surgical wound.
* the impact of postoperative hemoglobin (Hb) reduction on patients' quality of life.
* the impact of topical application of TA on the length of hospital stay.
* the impact of topical application of TA on ROM, pain, and surgical infection rate of the knee joint.
* the incidence of autologous and allogenic blood transfusion in patients receiving the standard.
* multimodal blood conservation techniques for TKA surgery at our institution
* to compare the efficacy and safety of high dose (3 g) of TA versus low dose (1.5 g) of TA.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (greater than 18 years old).
* Patients scheduled for primary unilateral total knee arthroplasty.

Exclusion Criteria:

* Allergy to tranexamic acid
* Acquired disturbances of color vision
* Preoperative anemia (hemoglobin <110 in females; hemoglobin <120 in males)
* Refusal of blood products (Jehovah's witnesses),
* Preoperative use of anticoagulant therapy - coumadin, heparin within 5 days of surgery, fibrinolytic disorders requiring intraoperative antifibrinolytic treatment,
* Coagulopathy (preoperative platelet count < 150,000/mm3, INR >1.4, prolonged PTT (>1.4 x normal))
* A previous history of thromboembolic disease (e.g. CVA, DVT or PE)
* Pregnancy
* Breastfeeding
* Significant co-morbidities:
* severe ischemic heart disease; NYHA Class III, IV,
* previous myocardial infarction
* severe pulmonary disease, e.g. FEV1<50% normal,
* plasma creatinine greater than 115 µmol/l in males and more than 100 µmol/l in females
* hepatic failure
* Intraoperative surgical/medical/anesthetic complications occur, e.g. MI, intraoperative bone fracture or neurovascular injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Calculated blood loss | Postoperative day 1-3

SECONDARY OUTCOMES:
Total prevalence of drug-related adverse events | one month after the medication/placebo administration
perioperative packed red blood cell transfusion requirements | Intraoperative and postoperative day 1-3
Systemic absorption of TA after topical application into the surgical wound | 1 hr after the surgey (after touniquet release)
length of hospital stay | postoperative
The change in the knee joint range of motion at flexion | Postoperative day 2
The amount of pain at the knee joint measured by a visual scale (VAS) | Postoperative week 6
Health-related quality of life determined by the Western Ontario and Mac Master Universities Osteoarthritis (WOMAC) index score | Postoperative week 6

CONTACTS AND LOCATIONS:
Overall Officials: Jean Wong, MD, FRCPC, Principal Investigator — Staff Anesthesiologist , Assistant Professor, Department of Anesthesia, Toronto Western Hospital
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada